CLINICAL TRIAL: NCT03574519
Title: Project Step II: The Effects of Incentives and Feedback on Promoting Walking Within Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Psi Chi (Other); Qualtrics (Unknown); American College of Sports Medicine (Other)
Responsible Party: Principal Investigator, Stephanie Kerrigan, Principal Investigator, Drexel University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1601004185-2
Record Dates: First submitted 2018-06-12; First posted 2018-07-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Physical Activity; Sedentary Lifestyle; Overweight and Obesity
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-contingent incentives and weekly feedback (Experimental): Participants will receive payment for participating in the study (regardless of goal attainment) and will receive weekly updates about their performance.
  Interventions: Behavioral: Non-contingent incentives; Behavioral: Weekly feedback
- Non-contingent incentives and daily feedback (Experimental): Participants will receive payment for participating in the study (regardless of goal attainment) and will receive daily updates about their performance.
  Interventions: Behavioral: Non-contingent incentives; Behavioral: Daily feedback
- Contingent incentives and weekly feedback (Experimental): Participants will receive payment for meeting their daily goals and will receive weekly updates about their performance.
  Interventions: Behavioral: Contingent incentives; Behavioral: Weekly feedback
- Contingent incentives and daily feedback (Experimental): Participants will receive payment for meeting their daily goals and will receive daily updates about their performance.
  Interventions: Behavioral: Contingent incentives; Behavioral: Daily feedback

INTERVENTIONS:
Behavioral: Non-contingent incentives — Incentives are provided for participation
  Arms: Non-contingent incentives and daily feedback; Non-contingent incentives and weekly feedback
Behavioral: Contingent incentives — Incentives are provided for attaining daily goals
  Arms: Contingent incentives and daily feedback; Contingent incentives and weekly feedback
Behavioral: Weekly feedback — Text message feedback is delivered weekly summarizing the past week's progress
  Arms: Contingent incentives and weekly feedback; Non-contingent incentives and weekly feedback
Behavioral: Daily feedback — Text message feedback is delivered daily summarizing the current day's progress
  Arms: Contingent incentives and daily feedback; Non-contingent incentives and daily feedback

SUMMARY:
This study will evaluate the main effects of daily vs. weekly feedback and contingent vs. non-contingent incentives for increasing walking behavior among overweight and obese adults.

DETAILED DESCRIPTION:
Approximately 68% of adults are overweight or obese, which is associated with increased risk for health conditions, including cardiovascular disease, type 2 diabetes, and cancer. These individuals are more often sedentary than the general population, which compounds the risk for these same conditions. While the benefits of engaging in physical activity are well-established, few individuals are able to successfully increase activity to recommended levels. Existing intervention programs, often derived from theories such as social cognitive theory or related theories, have had limited success. Behavioral economics offers a promising alternative, suggesting that engagement in any behavior is based on the maximizing utility and happiness (i.e., weighing the cost and benefit of the behavior). Interventions based on this theory aim to increase the immediate benefit of engaging in physical activity, often using a financial incentive.

This study will last for 8 weeks. All participants will have the use of a FitBit for ongoing self-monitoring and a personalized step-count goal designed to help increase daily steps. Participants will receive feedback on reaching their goals either daily or weekly.

ELIGIBILITY:
Inclusion Criteria:

* 25 kg/m2 ≤ BMI ≤ 45 kg/m2
* Age 18-70
* Currently inactive (engages in less than 6,000 steps/day on at least 4 of 7 days per week OR engaged in less than 10,000 steps /day on at least 5/7 days per week, confirmed by FitBit at baseline)
* Able to engage in moderate amount of walking
* Able to receive email/text messages from study staff

Exclusion Criteria:

* Psychiatric conditions that would make it difficult to comply
* Medical conditions that would make it difficult to comply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Step counts | Change from baseline to end of 6-week intervention
  Average daily step counts

SECONDARY OUTCOMES:
Step counts | Change from end of intervention to end of 2-week follow-up
  Average daily step counts
Step counts | Daily change during 6-week intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerrigan SG, Forman EM, Williams D, Patel M, Loyka C, Zhang F, Crosby RD, Butryn ML. Project Step: A Randomized Controlled Trial Investigating the Effects of Frequent Feedback and Contingent Incentives on Physical Activity. J Phys Act Health. 2021 Mar 1;18(3):247-253. doi: 10.1123/jpah.2020-0198. Epub 2021 Feb 17. PMID 33601334